CLINICAL TRIAL: NCT03127189
Title: A Phase 1, Open-label, Randomized, Parallel-group Study in Healthy Subjects to Investigate the Effect of Different Particle Sizes on the Single-dose Pharmacokinetics of Rilpivirine After Intramuscular Injection of a Long-acting Nanosuspension
Brief Title: A Study to Investigate the Effect of Different Particle Sizes on the Single-dose Pharmacokinetics of Rilpivirine After Intramuscular Injection of a Long-acting Nanosuspension in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108302; TMC278LAHTX1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-03-15; First posted 2017-04-25 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1-RPV LA: Treatment B (Experimental): Participants will receive single dose of 25 milligram (mg) rilpivirine (RPV) as an oral solution on Day 1 in Session 1 and Treatment B containing a single intramuscular (IM) injection of 600 mg rilpivirine long-acting parenteral formulation (RPV LA) [with different particle size distribution (PSD) as compared to Treatment A, D, C and E] on Day 1 of session 2. Both the sessions are separated by a wash-out Period of at least 14 days.
  Interventions: Drug: Rilpivirine; Drug: Rilpivirine Long-acting Parenteral Formulation
- Cohort 1-RPV LA: Treatment D (Experimental): Participants will receive single dose of 25 mg rilpivirine (RPV) as an oral solution on Day 1 in Session 1 and Treatment D containing a single IM injection of 600 mg RPV LA [with different PSD as compared to Treatment A, B, C and E) on Day 1 of session 2. Both the sessions are separated by a wash-out Period of at least 14 days.
  Interventions: Drug: Rilpivirine; Drug: Rilpivirine Long-acting Parenteral Formulation
- Cohort 2-RPV LA: Treatment A (Experimental): Participants will receive single dose of 25 mg rilpivirine (RPV) as an oral solution on Day 1 in Session 1 and Treatment A containing a single IM injection of 600 mg RPV LA [with different PSD as compared to Treatment B, C, D and E] on Day 1 of session 2. Both the sessions are separated by a wash-out Period of at least 14 days.
  Interventions: Drug: Rilpivirine; Drug: Rilpivirine Long-acting Parenteral Formulation
- Cohort 2-RPV LA: Treatment C (Experimental): Participants will receive single dose of 25 mg rilpivirine (RPV) as an oral solution on Day 1 in Session 1 and Treatment C containing a single IM injection of 600 mg RPV LA [with different PSD as compared to Treatment A, B, D and E] on Day 1 of session 2. Both the sessions are separated by a wash-out Period of at least 14 days.
  Interventions: Drug: Rilpivirine; Drug: Rilpivirine Long-acting Parenteral Formulation
- Cohort 2-RPV LA: Treatment E (Experimental): Participants will receive single dose of 25 mg rilpivirine (RPV) as an oral solution on Day 1 in Session 1 and Treatment E containing a single IM injection of 600 mg RPV LA [with different PSD as compared to Treatment A, B, C and D] on Day 1 of session 2. Both the sessions are separated by a wash-out Period of at least 14 days.
  Interventions: Drug: Rilpivirine; Drug: Rilpivirine Long-acting Parenteral Formulation

INTERVENTIONS:
Drug: Rilpivirine — Rilpivirine 25 mg immediate release oral solution.
Drug: Rilpivirine Long-acting Parenteral Formulation — RPV LA 600 mg extended-release suspension for IM injection.

SUMMARY:
The main purpose of this study is to characterize the single-dose pharmacokinetics (PK) of rilpivirine (RPV) after intramuscular (IM) injection of rilpivirine long-acting parenteral formulation (RPV LA) nanosuspensions with different particle size distribution (PSD), in healthy adult participants.

DETAILED DESCRIPTION:
This is a phase 1, open-label (all people know the identity of the intervention), randomized (study medication is assigned by chance), parallel-group, sequential study in healthy adult participants to characterize the single-dose pharmacokinetics (PK) of rilpivirine (RPV) after intramuscular (IM) injection of RPV LA nanosuspensions with different particle size distributions (PSD), in healthy adult participants. A total of 110 healthy adult participants will be enrolled in this study. The study will consist of 2 treatment sessions in a fixed sequential order: Session 1- all participants will receive a single oral dose of rilpivirine 25 milligram (mg) as oral immediate release solution on Day 1; Session 2- the participants will be randomized in session 2 on Day 1 in a 1:1:1:1:1 ratio to Treatments A, B, C, D and E. Each treatment group will receive a single IM injection of RPV LA on Day 1 of session 2. Session 1 and 2 will be separated by a washout period of at least 14 days. The total study duration for each participant will be approximately 9.5 months. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies
* A female participant of childbearing potential must have a negative serum beta-human chorionic gonadotropin test at screening and on Day -1 of each session
* For the duration of the study and for at least 6 months after intramuscular (IM) injection of rilpivirine long-acting parenteral formulation (RPV LA) (or 1 month after administration of rilpivirine (RPV) oral solution for participants who discontinue after Session 1), male and female participants must agree to practice effective methods of contraception, and must agree not to donate sperm (males)/eggs (ova, oocytes; for females) for the purposes of assisted reproduction
* Participant must be non-smoking for at least 3 months prior to screening

Exclusion Criteria:

* Female participant who is breastfeeding at screening
* Participant with a history of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant or that could prevent, limit or confound the protocol specified assessments. This may include, but is not limited to, renal dysfunction, significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* Participant has a history of clinically relevant arrhythmias or history of risk factors for Torsade de Pointes (hypokalemia, family history of long QT)
* Participant has clinically relevant, currently active, or underlying gastrointestinal, cardiovascular, nervous system, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory or infectious disease
* Participant has known allergies, hypersensitivity, or intolerance to RPV or its excipients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Session 2: Maximum Observed Plasma Concentration (Cmax) | Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 408, 528, 672, 1344, 2016, 2688, 3360, 4032, 4704, 5376, and 6048 hours post-dose
  The Cmax is the maximum observed plasma concentration.
Session 2: Area Under the Plasma Concentration-Time Curve From Time Zero (Day 1) to Day 28 (AUC[0-d28]) | 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 408, and 528 hours post-dose
  The AUC (0-d28) is the area under the plasma concentration-time curve from time of administration up to Day 28 postdose.
Session 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 408, 528, 672, 1344, 2016, 2688, 3360, 4032, 4704, 5376, and 6048 hours post-dose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Session 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168,216, 264, 336, 408, 528, 672, 1344, 2016, 2688, 3360, 4032, 4704, 5376, and 6048 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Baseline, up to 9.5 months
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Session 1: Maximum Observed Plasma Concentration (Cmax) | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120 and 168 hours post-dose
  The Cmax is the maximum observed plasma concentration.
Session 1: Area Under the Plasma Concentration-Time Curve From Time Zero (Day 1) to Day 28 AUC (0-d28) | 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120, 168, hours post-dose
  The AUC (0-d28) is the area under the plasma concentration time curve from time of administration up to Day 28 postdose.
Session 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time AUC (0-last) | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120 and 168 hours post-dose
  The AUC (0-last) is the area under the plasma concentration time curve from time zero to last quantifiable time.
Session 1: Area Under the Plasma Concentration-Time Curve From Time Zero To Infinite Time AUC (0-infinity) | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120 and 168 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z). wherein AUC(last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Celerion, Tempe, Arizona
  - Celerion, Lincoln, Nebraska